CLINICAL TRIAL: NCT05883748
Title: HELIOS: An Open-Label, Long-Term Study to Investigate the Safety, Tolerability, and Efficacy of DISC-1459 (Bitopertin) in Participants With Erythropoietic Protoporphyria (EPP) or X-Linked Protoporphyria (XLP)
Brief Title: HELIOS: Open-Label, Long-Term Extension Study to Investigate the Safety, Tolerability, and Efficacy of DISC-1459 (Bitopertin) in Participants With EPP or XLP
Status: Enrolling by invitation | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Disc Medicine, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DISC-1459-501
Record Dates: First submitted 2023-05-22; First posted 2023-06-01 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Erythropoietic Protoporphyria
Keywords: EPP; DISC-1459; porphyria; RO4917838
MeSH Terms: conditions — Protoporphyria, Erythropoietic; Porphyrias | interventions — (4-(3-fluoro-5-trifluoromethylpyridin-2-yl)piperazin-1-yl)(5-methanesulfonyl-2-(2,2,2-trifluoro-1-methylethoxy)phenyl)methanone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- DISC-1459 Oral Dose Level 1 (Experimental): Oral dose, once a day
  Interventions: Drug: DISC-1459
- DISC-1459 Oral Dose Level 2 (Experimental): Oral dose, once a day
  Interventions: Drug: DISC-1459

INTERVENTIONS:
Drug: DISC-1459 — DISC-1459 dose level 1
  Other Names: Bitopertin; RO4917838
  Arms: DISC-1459 Oral Dose Level 1
Drug: DISC-1459 — DISC-1459 dose level 2
  Other Names: Bitopertin; RO4917838
  Arms: DISC-1459 Oral Dose Level 2

SUMMARY:
This is an open-label, long-term extension study to investigate the safety, tolerability and efficacy of DISC-1459 in participants with EPP.

ELIGIBILITY:
Inclusion Criteria:

* Participants with diagnosis of EPP who are participating (or who have participated) in a prior Disc Medicine bitopertin study and who have completed the randomized treatment phase and End-of-Study visit
* Aged ≥12 years upon study consent
* Body weight ≥32 kg for participants <18 years of age and BMI ≥18.5 kg/m2 for adult participants
* Willing to practice highly effective methods of birth control (both males who have partners of childbearing potential and females of childbearing potential during the study, while taking study drug, and for at least 30 days after the last dose of study drug.
* Negative urine or serum pregnancy test (females of childbearing potential).
* Able to understand the study aims, procedures, and requirements, and provide written informed consent (and assent if necessary).
* Able to comply with all study procedures.

Exclusion Criteria:

* Participants who have an ongoing SAE from a clinical study that is assessed by the investigator as related to bitopertin
* Other medical or psychiatric condition or laboratory finding not specifically noted above that, in the judgement of the Investigator or Sponsor, would put the participant at unacceptable risk or otherwise preclude participation in the study
* Condition or concomitant medication that would confound the ability to interpret clinical, clinical laboratory, or participant diary data, including a major psychiatric condition that has had an exacerbation or required hospitalization in the last 6 months
* Planned treatment with afamelanotide or dersimelagon during the study
* Planned use of any drugs or herbal remedies known to be strong inhibitors or inducers of cytochrome p450 (CYP)3A4 enzymes throughout the study
* If female, pregnant, or breastfeeding
* Participation in any other clinical protocol or investigational trial, other than Disc Medicine bitopertin trials, that involves administration of experimental therapy and/or therapeutic devices within 30 days of Day 1
* Score of PHQ-8 ≥10 at screening or imminent suicidal risk identified by the C-SSRS as defined as suicidal ideation with intent (Grade 4 or 5) within the last year or any suicidal behavior within the last 5 years.
* Consumption of grapefruit/Seville orange and products containing these for 14 days prior to first dose of study drug and throughout the study

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2023-08-31 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events | up to 5 Years
Incidence of clinically abnormal vital signs | up to 5 Years
Incidence of clinically abnormal physical exam | up to 5 Years
Incidence of abnormal laboratory test results | up to 5 Years
Assessment of Patient Health Questionnaire (PHQ-8) | up to 5 Years
  The Patient Health Questionnaire (PHQ-8), an 8-item participant-report measure for screening for depression and for establishing depression severity. The total score ranges from 0-24, with a higher score indicating greater depression symptom severity.
Assessment of C-SSRS | up to 5 Years
  The C-SSRS is a clinician-rated scale that assesses suicidality from ideation to behaviors and monitors the potential emergence of suicidality in clinical studies.

SECONDARY OUTCOMES:
Change from baseline in daily daylight tolerance, as assessed by total hours spent in the sunlight without pain and average time to first prodromal syndrome in sunlight | up to 5 Years
Change from baseline in whole blood metal-free PPIX levels | up to 5 Years
Plasma Bitopertin Concentrations | up to 5 Years

CONTACTS AND LOCATIONS:
Overall Officials: Will Savage, MD PhD, Study Director — Disc Medicine
Locations (13):
- United States (11):
  - University of Alabama Hospital, Birmingham, Alabama
  - University of California San Francisco, San Francisco, California
  - University of Miami Miller School of Medicine, Miami, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - MetroBoston Clinical Partners, Boston, Massachusetts
  - Mount Sinai Hospital, New York, New York
  - Atrium Health Wake Forest Baptist, Winston-Salem, North Carolina
  - Remington-Davis Clinical Research, Columbus, Ohio
  - Einstein Medical Center, Philadelphia, Pennsylvania
  - University of Texas, Galveston, Texas
  - Fred Hutchinson Cancer Center, Seattle, Washington
- Australia (2):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - The Royal Melbourne Hospital, Parkville, Victoria

IPD SHARING:
Plan to Share IPD: No